CLINICAL TRIAL: NCT00507026
Title: Randomized, Double-Blind, Active-and Placebo-Controlled Study of the Analgesic Efficacy and Safety of Repeated Dosing of DIC075V Versus Parenteral Ketorolac and Placebo in Acute Post-Operative Pain After Elective Orthopedic Surgery
Brief Title: Efficacy and Safety of IV Diclofenac (DIV075V)for Pain After Elective Orthopedic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFC-005; C1211009 (Other: Alias Study Number)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- A (Experimental): DIC075V (IV diclofenac)
  Interventions: Drug: IV Diclofenac
- B (Active Comparator): IV Ketorolac
  Interventions: Drug: IV ketorolac
- C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Diclofenac — IV Diclofenac q6h
  Arms: A
Drug: IV ketorolac — IV ketorolac q6h
  Arms: B
Drug: Placebo — Placebo q6h
  Arms: C

SUMMARY:
This study will compare repeated intermittent IV dosing of diclofenac in patient with moderate to severe post-surgical pain from elective orthopedic surgery.

DETAILED DESCRIPTION:
The primary objective is to evaluate the analgesic efficacy and safety of three dosage levels of parenteral diclofenac in providing pain relief as compared to placebo or Ketorolac tromethamine.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled within three weeks of the screening visit to undergo elective orthopedic surgery.
* Moderate to severe pain within 6 hours following completion of the required surgery.

Exclusion Criteria:

* Chronic pain conditions.
* Chronic disease or recent cardiovascular events.
* Known allergy or hypersensitivity to the active compounds or any of the excipients used in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2007-07-25 (Actual); Primary Completion 2008-10-14 (Actual); Study Completion 2008-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Helen Keller Hospital, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Accurate Clinical Trials, San Clemente, California
  - East Coast Clincial Research, Ft. Pierce, Florida
  - Outcomes Research Institute, Louisville, Kentucky
  - American Institute of Healthcare and Fitness, Raleigh, North Carolina
  - University Orthopedics Center, State College, Pennsylvania
  - SCIREX, Austin, Texas

REFERENCES:
- [Derived] Chelly JE, Lacouture PG, Reyes CRD. Safety of Injectable HPbetaCD-Diclofenac in Older Patients with Acute Moderate-to-Severe Postoperative Pain: A Pooled Analysis of Three Phase III Trials. Drugs Aging. 2018 Mar;35(3):249-259. doi: 10.1007/s40266-018-0529-3. PMID 29492863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who required elective general orthopedic surgery were eligible for participation in this study. Within 6 hours after completion of surgery, participants who experienced moderate to severe pain, as measured by a 0-100 millimeter (mm) visual analog scale (VAS) with pain intensity (PI) score of greater than or equal to (>=) 50 mm and who met all eligibility criteria were enrolled into the study.
Pre-assignment Details: Total 432 participants signed the inform consent form (ICF). Out of which 155 participants were not admitted into the study, 277 actually enrolled into the study and assigned to study treatment.
Groups:
- Diclofenac (DIC075V): Participants at high risk (weighing less than [<] 50 killogram [k]), age >= 65 years, elevated nonsteroidal anti-inflammatory drugs [NSAID]-related gastrointestinal [GI] risk factors, or with hepatic or renal impairment) received DIC075V 18.75 milligram (mg). Participants without any risk factor and weighing greater than (>) 95 kg received DIC075V 50 mg. Participants weighing >95 kg with any risk factor received DIC075V 18.75 mg. All other participants received DIC075V 37.5 mg. DIC075V was administered as intravenous (IV) bolus every 6 hours for up to 5 days. Participants returned to the clinic for a safety follow-up 5-9 days after discharge and had a safety follow-up telephone call 30-37 days after the last study drug administration.
- Ketorolac: Participants at high risk (weighing <50 k, >=65 years, elevated NSAID-related GI risk factors, or with hepatic or renal impairment) received ketorolac tromethamine 15 mg. Participants without any risk factor and weighing >95 kg received ketorolac tromethamine 30 mg. Participants weighing >95 kg with any risk factor received ketorolac tromethamine 15 mg. All other participants received ketorolac tromethamine 30 mg. Ketorolac tromethamine was administered as IV bolus every 6 hours for up to 5 days. Participants returned to the clinic for a safety follow-up 5-9 days after discharge and had a safety follow-up telephone call 30-37 days after the last study drug administration.
- Placebo: Participants received saline as placebo as IV bolus every 6 hours for up to 5 days. Participants returned to the clinic for a safety follow-up 5-9 days after discharge and had a safety follow-up telephone call 30-37 days after the last study drug administration.
Period: Overall Study
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Started | 145 | 60 | 72
Completed | 132 | 56 | 51
Not Completed | 13 | 4 | 21
Not completed — Lack of Efficacy | 6 | 4 | 21
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Investigator Decision | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population included all participants who were randomized into the study and who received at least 1 dose of study medication.
Groups:
- Diclofenac (DIC075V): Participants at high risk (weighing <50 k), age >= 65 years, elevated NSAID-related GI risk factors, or with hepatic or renal impairment) received DIC075V 18.75 mg. Participants without any risk factor and weighing >95 kg received DIC075V 50 mg. Participants weighing >95 kg with any risk factor received DIC075V 18.75 mg. All other participants received DIC075V 37.5 mg. DIC075V was administered as IV bolus every 6 hours for up to 5 days. Participants returned to the clinic for a safety follow-up 5-9 days after discharge and had a safety follow-up telephone call 30-37 days after the last study drug administration.
- Total: Total of all reporting groups
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo | Total
Number analyzed (Participants) | 145 | 60 | 72 | 277
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (14.35) | 54.9 (15.77) | 54.5 (15.67) | 55.3 (14.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 40 | 46 | 178
  Male | 53 | 20 | 26 | 99

OUTCOME MEASURES:

1. Primary Outcome: Sum of the Pain Intensity Differences (SPID) Over 24 Hours
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. SPIDs was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 24 hours ranges from -2400 to 2400. A higher value indicates a better pain reduction.
Time Frame: Over 24 hours post first dose
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours | 577.0 (570.90) | 563.2 (586.21) | 28.0 (428.43)
Statistical Analysis 1: Comparison: Diclofenac (DIC075V) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Ketorolac vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

2. Primary Outcome: Sum of the Pain Intensity Differences (SPID) Over 48 Hours
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, PID is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. SPIDs was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 48 hours ranges from -4800 to 4800. A higher value indicates a better pain reduction.
Time Frame: Over 48 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours | 1527.5 (1139.30) | 1371.8 (1152.19) | 400.4 (949.54)
Statistical Analysis 1: Comparison: Diclofenac (DIC075V) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Ketorolac vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

3. Primary Outcome: Sum of the Pain Intensity Differences (SPID) Over 72 Hours
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, PID is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. SPIDs was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 72 hours ranges from -7200 to 7200. A higher value indicates a better pain reduction.
Time Frame: Over 72 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours | 2592.1 (1730.92) | 2312.1 (1743.73) | 836.8 (1564.24)
Statistical Analysis 1: Comparison: Diclofenac (DIC075V) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Ketorolac vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

4. Primary Outcome: Sum of the Pain Intensity Differences (SPID) Over 96 Hours
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, PID is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. SPIDs was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 96 hours ranges from -9600 to 9600. A higher value indicates a better pain reduction.
Time Frame: Over 96 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours | 3711.3 (2347.25) | 3331.9 (2356.36) | 1337.8 (2261.50)
Statistical Analysis 1: Comparison: Diclofenac (DIC075V) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Ketorolac vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

5. Primary Outcome: Sum of the Pain Intensity Differences (SPID) Over 120 Hours
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, PID is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. SPIDs was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 120 hours ranges from -12000 to 12000. A higher value indicates a better pain reduction.
Time Frame: Over 120 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours | 4835.6 (2988.78) | 4359.1 (3001.32) | 1840.5 (2987.85)
Statistical Analysis 1: Comparison: Diclofenac (DIC075V) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Ketorolac vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

6. Secondary Outcome: Pain Intensity Differences (PID) Over Time
Description: Pain intensity was measured on VAS (from 0 mm to 100 mm: 0 = no pain, 100 = worst possible pain). For each post dose time point, PID is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). PID score range at any post dose (post baseline) evaluation time point was -100 to 100. A positive difference score is indicative of improvement.
Time Frame: Baseline (0 hour), 5, 10, 15, 30, 45 minutes post first dose, 1, 2, 3, 5, 6, 9, 12, 15, 18, 21, 24, 48, 72, 96, 120 hours post first dose
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 144 | 60 | 71
mm
  At 5 minutes | 5.2 (14.27) | 3.2 (15.85) | 1.2 (15.21)
  At 10 minutes: number analyzed (Participants) | 143 | 60 | 71
  At 10 minutes | 9.1 (19.36) | 5.5 (19.61) | 2.4 (21.46)
  At 15 minutes: number analyzed (Participants) | 142 | 59 | 69
  At 15 minutes | 13.4 (22.06) | 9.8 (23.21) | 2.2 (25.41)
  At 30 minutes: number analyzed (Participants) | 134 | 53 | 59
  At 30 minutes | 17.7 (24.36) | 16.7 (23.22) | 2.6 (30.16)
  At 45 minutes: number analyzed (Participants) | 115 | 45 | 37
  At 45 minutes | 18.5 (27.12) | 18.4 (27.56) | -1.2 (30.15)
  At 1 hour: number analyzed (Participants) | 107 | 40 | 32
  At 1 hour | 18.7 (28.54) | 19.7 (31.60) | -4.2 (28.03)
  At 2 hours: number analyzed (Participants) | 82 | 31 | 16
  At 2 hours | 17.3 (30.22) | 16.9 (32.81) | -7.8 (23.86)
  At 3 hours: number analyzed (Participants) | 76 | 27 | 13
  At 3 hours | 13.5 (29.30) | 14.7 (32.94) | -8.9 (19.21)
  At 5 hours: number analyzed (Participants) | 72 | 31 | 10
  At 5 hours | 10.8 (30.11) | 15.1 (32.01) | -7.3 (20.76)
  At 6 hours: number analyzed (Participants) | 81 | 33 | 16
  At 6 hours | 12.6 (31.05) | 12.5 (29.69) | -6.1 (21.31)
  At 9 hours: number analyzed (Participants) | 76 | 29 | 14
  At 9 hours | 23.6 (32.07) | 21.3 (33.34) | -1.8 (22.91)
  At 12 hours: number analyzed (Participants) | 103 | 38 | 28
  At 12 hours | 23.4 (31.83) | 23.7 (32.44) | 1.4 (24.75)
  At 15 hours: number analyzed (Participants) | 59 | 19 | 13
  At 15 hours | 28.5 (31.34) | 23.2 (35.19) | 1.1 (25.35)
  At 18 hours: number analyzed (Participants) | 109 | 45 | 35
  At 18 hours | 30.2 (32.27) | 30.1 (32.80) | 8.7 (24.16)
  At 21 hours: number analyzed (Participants) | 107 | 45 | 24
  At 21 hours | 36.3 (31.03) | 39.1 (32.41) | 8.8 (26.66)
  At 24 hours: number analyzed (Participants) | 102 | 41 | 30
  At 24 hours | 31.8 (32.47) | 27.5 (32.96) | 12.9 (26.38)
  At 48 hours: number analyzed (Participants) | 55 | 22 | 16
  At 48 hours | 42.9 (29.17) | 35.5 (30.38) | 19.4 (29.69)
  At 72 hours: number analyzed (Participants) | 17 | 4 | 2
  At 72 hours | 47.0 (27.65) | 41.0 (30.40) | 20.3 (31.44)
  At 96 hours: number analyzed (Participants) | 1 | 1 | 0
  At 96 hours | 46.8 (28.42) | 43.0 (28.92) |
  At 120 hours: number analyzed (Participants) | 67 | 25 | 19
  At 120 hours | 46.9 (28.42) | 42.9 (28.91) | 20.9 (31.48)

7. Secondary Outcome: Percentage of Participants Attaining Greater Than or Equal to (>=) 30 Percent (%) Reduction From Baseline in Pain Intensity
Description: Pain intensity was measured on a 0 to 100 mm VAS, larger values indicate greater pain intensity. In this outcome measure, percentage of participants attaining >= 30 % reduction in pain intensity from baseline to specified time points was reported.
Time Frame: Baseline (0 hour), 5, 30 minutes post first dose, 1, 24, 48, 72, 90, 120 hours post first dose
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
Percentage of participants
  At 5 minutes | 13.8 | 10.0 | 8.3
  At 30 minutes | 43.4 | 35.0 | 25.0
  At 1 hour | 44.8 | 41.7 | 15.3
  At 24 hours | 62.1 | 56.7 | 31.09
  At 48 hours | 75.2 | 63.3 | 41.7
  At 72 hours | 80.0 | 71.7 | 41.7
  At 90 hours | 80.0 | 75.0 | 43.1
  At 120 hours | 80.7 | 75.0 | 43.1

8. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: Pain relief values at specified time points were measured on a 0 to 100 mm VAS, where higher values indicate greater pain relief. TOTPAR over specified time interval was calculated as area under pain relief curve over specified time intervals using trapezoidal approximation. For 0-24 hours score range was 0-2400, for 0-48 hours score range was 0- 4800, for 0-96 hours score range was 0-9600 and for 0-120 hours score range was 0-12000. Higher TOTPAR values indicated more relief.
Time Frame: 0-24, 0-48, 0-72, 0-96 and 0-120 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*hours
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm*hours
  0-24 hours | 1177.6 (611.13) | 1065.4 (616.28) | 484.7 (502.91)
  0-48 hours | 2768.3 (1239.29) | 2453.8 (1323.35) | 1327.9 (1258.96)
  0-72 hours | 4471.0 (1898.89) | 3983.6 (2056.63) | 2214.6 (2103.25)
  0-96 hours | 6252.2 (2577.46) | 5575.7 (2828.49) | 3159.4 (3002.62)
  0-120 hours | 8042.5 (3282.39) | 7178.0 (3627.97) | 4105.4 (3922.22)

9. Secondary Outcome: Visual Analog Pain Relief Values Over the Time
Description: Pain relief values at specified time points were measured on a 0 to 100 mm VAS, where higher values indicate greater pain relief.
Time Frame: 5, 10, 15, 30, 45 minutes post first dose, 1, 2, 3, 5, 6, 9, 12, 15, 18, 21, 24, 48, 72, 96, 120 hours post first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
mm
  At 5 minutes | 21.9 (25.27) | 17.9 (25.26) | 15.3 (21.68)
  At 10 minutes | 27.1 (26.89) | 23.6 (28.15) | 19.0 (24.27)
  At 15 minutes | 33.5 (28.04) | 27.2 (30.74) | 21.6 (28.54)
  At 30 minutes | 39.7 (30.47) | 33.9 (33.04) | 23.1 (31.95)
  At 45 minutes | 41.6 (33.14) | 33.3 (33.64) | 19.9 (31.67)
  At 1 hour | 40.0 (34.64) | 37.8 (37.21) | 17.1 (30.67)
  At 2 hours | 35.3 (36.99) | 33.2 (37.98) | 10.1 (23.97)
  At 3 hours | 33.5 (37.06) | 29.5 (37.09) | 8.0 (22.07)
  At 5 hours | 28.8 (35.45) | 31.0 (36.74) | 8.0 (21.96)
  At 6 hours | 36.7 (34.78) | 33.9 (32.54) | 12.6 (24.10)
  At 9 hours | 49.5 (35.12) | 39.4 (34.59) | 17.5 (26.20)
  At 12 hours | 51.6 (33.42) | 46.3 (34.44) | 21.6 (27.46)
  At 15 hours | 55.7 (33.55) | 45.9 (34.08) | 21.4 (26.15)
  At 18 hours | 56.6 (33.00) | 53.6 (33.98) | 28.3 (30.07)
  At 21 hours | 63.6 (32.75) | 63.2 (33.05) | 27.4 (32.73)
  At 24 hours | 59.7 (33.73) | 53.4 (34.87) | 32.5 (35.25)
  At 48 hours | 69.4 (31.52) | 60.8 (33.83) | 38.2 (37.73)
  At 72 hours | 74.4 (31.01) | 64.8 (35.41) | 38.8 (38.77)
  At 96 hours | 74.6 (31.11) | 67.0 (34.96) | 39.4 (39.19)
  At 120 hours | 74.6 (31.15) | 66.9 (34.89) | 39.4 (39.19)

10. Secondary Outcome: Time From Administration of Study Drug to Administration of Rescue Medication
Description: Time from administration of study drug to administration of rescue medication were censored at time of last pain assessment for participants who did not receive rescue medication. Rescue medication was additional pain medication, available to participants if they did not receive pain relief from the study drug. Rescue medication available during this study was IV morphine.
Time Frame: Maximum up to 5 days
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication. Missing data was imputed using worst observation carried forward (WOCF) recorded over prior six hours (including baseline, if appropriate) in this outcome measure.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
Minutes | 220.0 [125.0 to 272.0] | 137.0 [63.0 to 302.0] | 51.0 [35.0 to 71.0]

11. Secondary Outcome: Cumulative Amount of Rescue Medication
Description: In this outcome measure, cumulative amount of rescue medication used over 0-24, 0-48, 0-72, 0-96, and 0-120 hours were reported. Rescue medication was additional pain medication, available to participants if they did not receive pain relief from the study drug. Rescue medication available during this study was IV morphine.
Time Frame: 0-24, 0-48, 0-72, 0-96 and 0-120 hours
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific rows. Missing data was imputed using WOCF recorded over prior six hours (including baseline, if appropriate) in this outcome measure.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 107 | 44 | 68
mg
  0-24 hours: number analyzed (Participants) | 106 | 43 | 68
  0-24 hours | 9.4 (7.20) | 11.5 (7.81) | 16.0 (10.61)
  0-48 hours | 11.1 (9.06) | 15.5 (13.99) | 19.0 (13.89)
  0-72 hours | 11.7 (9.56) | 18.0 (20.11) | 20.5 (16.19)
  0-96 hours | 11.8 (9.73) | 18.1 (20.14) | 20.5 (16.17)
  0-120 hours | 11.8 (9.73) | 18.1 (20.17) | 20.5 (16.17)

12. Secondary Outcome: Number of Participants According to Frequency of Use of Rescue Medication
Description: In this outcome measure, number of participants are reported according to number of times they received rescue medication. Rescue medication was additional pain medication, available to participants if they did not receive pain relief from the study drug. Rescue medication available during this study was IV morphine. Only those categories with at least one nonzero value are reported.
Time Frame: 0-24, 0-48, 0-72, 0-96 and 0-120 hours post first dose
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication. Missing data was imputed using WOCF recorded over prior six hours (including baseline, if appropriate) in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
Participants
  0 - 24 Hours: 0 | 39 | 17 | 4
  0 - 24 Hours: 1 | 26 | 6 | 7
  0 - 24 Hours: 2 | 26 | 9 | 6
  0 - 24 Hours: 3 | 19 | 8 | 11
  0 - 24 Hours: 4 | 8 | 4 | 9
  0 - 24 Hours: 5 | 9 | 3 | 9
  0 - 24 Hours: 6 | 7 | 3 | 3
  0 - 24 Hours: 7 | 3 | 5 | 7
  0 - 24 Hours: 8 | 2 | 2 | 4
  0 - 24 Hours: 9 | 3 | 1 | 4
  0 - 24 Hours: 11 | 1 | 1 | 3
  0 - 24 Hours: 12 | 1 | 1 | 2
  0 - 24 Hours: 13 | 1 | 0 | 1
  0 - 24 Hours: 14 | 0 | 0 | 1
  0 - 24 Hours: 15 | 0 | 0 | 1
  0-48 hours: 0 | 38 | 16 | 14
  0-48 hours: 1 | 23 | 5 | 7
  0-48 hours: 2 | 24 | 10 | 6
  0-48 hours: 3 | 14 | 5 | 10
  0-48 hours: 4 | 11 | 2 | 3
  0-48 hours: 5 | 7 | 3 | 8
  0-48 hours: 6 | 8 | 2 | 5
  0-48 hours: 7 | 6 | 4 | 8
  0-48 hours: 8 | 3 | 3 | 3
  0-48 hours: 9 | 4 | 4 | 5
  0-48 hours: 10 | 2 | 2 | 0
  0-48 hours: 11 | 3 | 1 | 5
  0-48 hours: 12 | 1 | 2 | 3
  0-48 hours: 13 | 1 | 1 | 1
  0-48 hours: 14 | 0 | 0 | 1
  0-48 hours: 15 | 0 | 0 | 1
  0-48 hours: 17 | 0 | 0 | 1
  0-48 hours: 20 | 0 | 0 | 1
  0-72 hours: 0 | 38 | 16 | 4
  0-72 hours: 1 | 23 | 5 | 7
  0-72 hours: 2 | 22 | 10 | 6
  0-72 hours: 3 | 15 | 5 | 10
  0-72 hours: 4 | 11 | 2 | 3
  0-72 hours: 5 | 6 | 2 | 5
  0-72 hours: 6 | 8 | 2 | 7
  0-72 hours: 7 | 4 | 4 | 6
  0-72 hours: 8 | 4 | 2 | 2
  0-72 hours: 9 | 3 | 1 | 9
  0-72 hours: 10 | 5 | 4 | 9
  0-72 hours: 11 | 3 | 2 | 0
  0-72 hours: 12 | 2 | 1 | 2
  0-72 hours: 13 | 1 | 1 | 3
  0-72 hours: 14 | 0 | 0 | 1
  0-72 hours: 15 | 0 | 2 | 2
  0-72 hours: 17 | 0 | 1 | 0
  0-72 hours: 19 | 0 | 0 | 1
  0-72 hours: 20 | 0 | 0 | 1
  0-72 hours: 21 | 0 | 0 | 1
  0-96 hours: 0 | 38 | 16 | 4
  0-96 hours: 1 | 23 | 5 | 7
  0-96 hours: 2 | 22 | 10 | 6
  0-96 hours: 3 | 15 | 5 | 10
  0-96 hours: 4 | 11 | 2 | 3
  0-96 hours: 5 | 6 | 2 | 5
  0-96 hours: 6 | 7 | 2 | 6
  0-96 hours: 7 | 5 | 4 | 7
  0-96 hours: 8 | 3 | 2 | 2
  0-96 hours: 9 | 3 | 1 | 9
  0-96 hours: 10 | 5 | 3 | 0
  0-96 hours: 11 | 3 | 3 | 2
  0-96 hours: 12 | 3 | 1 | 3
  0-96 hours: 13 | 1 | 1 | 1
  0-96 hours: 14 | 0 | 0 | 2
  0-96 hours: 15 | 0 | 2 | 2
  0-96 hours: 17 | 0 | 1 | 0
  0-96 hours: 19 | 0 | 0 | 1
  0-96 hours: 20 | 0 | 0 | 1
  0-96 hours: 21 | 0 | 0 | 1
  0-120 hours: 0 | 38 | 16 | 4
  0-120 hours: 1 | 23 | 5 | 7
  0-120 hours: 2 | 22 | 10 | 6
  0-120 hours: 3 | 15 | 5 | 10
  0-120 hours: 4 | 11 | 2 | 3
  0-120 hours: 5 | 6 | 2 | 5
  0-120 hours: 6 | 7 | 2 | 6
  0-120 hours: 7 | 5 | 4 | 7
  0-120 hours: 8 | 3 | 2 | 2
  0-120 hours: 9 | 3 | 1 | 9
  0-120 hours: 10 | 5 | 3 | 0
  0-120 hours: 11 | 3 | 2 | 2
  0-120 hours: 12 | 3 | 2 | 3
  0-120 hours: 13 | 1 | 1 | 1
  0-120 hours: 14 | 0 | 0 | 2
  0-120 hours: 15 | 0 | 2 | 2
  0-120 hours: 17 | 0 | 1 | 0
  0-120 hours: 19 | 0 | 0 | 1
  0-120 hours: 20 | 0 | 0 | 1
  0-120 hours: 21 | 0 | 0 | 1

13. Secondary Outcome: Participant Global Evaluation Over Time
Description: Participants global evaluation of study medication was accessed on a scale ranging from scale 0 to 4 where 0= poor, 1= fair, 2= good, 3= very good, 4= excellent where higher score represented better outcome.
Time Frame: 0-24, 0-48, 0-120 hours post-dose
Population: ITT population included all participants who were randomized into the study and who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 141 | 59 | 70
Units on a scale
  0-24 Hours | 2.6 (1.27) | 2.4 (1.16) | 1.1 (1.25)
  0-48 Hours: number analyzed (Participants) | 60 | 26 | 20
  0-48 Hours | 2.9 (1.15) | 2.6 (0.86) | 1.9 (1.42)
  0-120 Hours | 2.9 (1.26) | 2.6 (1.16) | 1.3 (1.38)

14. Secondary Outcome: Time to Perceptible Relief
Description: Participants were instructed to stop the first stopwatch at the onset of perceptible pain relief after first dose. Event times of participants not reporting perceptible relief were censored at 6 hours; event times of participants who withdrew or were administered rescue medication were censored at time of withdrawal or rescue. Kaplan-Meier estimate was used for analysis.
Time Frame: Within 6 hours of first dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
Minutes | 10.0 [0 to 194] | 14.4 [0 to 85] | 15.0 [1 to 187]

15. Secondary Outcome: Time to Meaningful Relief
Description: Participants were instructed to stop the second stopwatch at the onset of meaningful pain relief after first dose. Event times of participants not reporting meaningful relief were censored at 6 hours; event times of participants who withdrew or were administered rescue medication were censored at time of withdrawal or rescue. Kaplan-Meier estimate was used for analysis.
Time Frame: Within 6 hours of first dose on Day 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Number analyzed (Participants) | 145 | 60 | 72
Minutes | 41.6 [31.0 to 58.6] | 42.5 [30.0 to 51.7] | NA [NA to NA] — Median and 95 % CI were not estimable as majority of participants in placebo arm did not achieve meaningful relief by 6 hours.

ADVERSE EVENTS:
Description: Same event may appear as both an adverse events (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Diclofenac (DIC075V) | Ketorolac | Placebo
Serious Adverse Events (participants affected / at risk) | 7/145 | 4/60 | 3/72
Other Adverse Events (participants affected / at risk) | 109/145 | 46/60 | 60/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac (DIC075V) (N=145) | Ketorolac (N=60) | Placebo (N=72)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac (DIC075V) (N=145) | Ketorolac (N=60) | Placebo (N=72)
Anaemia (Blood and lymphatic system disorders) | 9 | 7 | 8
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Eye oedema (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 19 | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 4 | 1 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 36 | 18 | 26
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 6 | 14
Adverse drug reaction (General disorders) | 0 | 1 | 0
Application site inflammation (General disorders) | 1 | 0 | 0
Application site reaction (General disorders) | 0 | 1 | 0
Application site vesicles (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Feeling drunk (General disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Infusion site erythema (General disorders) | 0 | 0 | 2
Infusion site pain (General disorders) | 11 | 5 | 5
Infusion site pruritus (General disorders) | 2 | 0 | 0
Infusion site reaction (General disorders) | 1 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Oedema peripheral (General disorders) | 8 | 3 | 2
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 3 | 9
Tenderness (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 8 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 7 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Incision site complication (Injury, poisoning and procedural complications) | 2 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 2 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 8 | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 3
Blood amylase increased (Investigations) | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 21 | 8 | 9
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1
Body temperature increased (Investigations) | 2 | 2 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 3
Haematocrit decreased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Confusional state (Nervous system disorders) | 1 | 0 | 2
Disorientation (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 16 | 5 | 5
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 12 | 5 | 5
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 7 | 4 | 5
Nightmare (Psychiatric disorders) | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 6 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 6 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.